CLINICAL TRIAL: NCT02200393
Title: Feasibility Study Using Abdominal Functional Electrical Stimulation (AFES) to Assist Ventilator Weaning in Tetraplegia
Brief Title: Abdominal Functional Electrical Stimulation (AFES) to Assist Ventilator Weaning in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Henrik Gollee, Senior Lecturer, University of Glasgow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN11NE458
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury; Tetraplegia
Keywords: Spinal cord injury; Tetraplegia; Ventilator
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abdominal FES (Experimental): Participants in the Abdominal Functional Electrical Stimulation (AFES) group will receive AFES 5 times per week (20 to 40 mins per day), on four alternate weeks.
  Interventions: Device: Abdominal FES

INTERVENTIONS:
Device: Abdominal FES — Stimulation intensity was adjusted on a channel by channel basis until a strong visible contraction of the abdominal muscles is observed. During the session, manual adjustment of both the stimulation intensity (to compensate for fatigue) and the duty cycle is possible.
  Four pairs of surface electrodes were placed on the participant's abdomen. One pair will be placed on both the right and left side of the rectus abdominis around the naval. One pair of electrodes will also be placed on both the right and left side of the external oblique muscles with one electrode being placed just below the participant's bottom rib and the other below this with a separation of around 3cm.
  Other Names: AFES; RehaStim

SUMMARY:
Compromised respiratory function as a result of tetraplegia leads to many tetraplegics requiring mechanical ventilation during the acute phase of injury. Mechanical ventilation is associated with additional costs to the local health care provider and reduced quality of life of the patient. Electrical stimulation of the abdominal muscles has previously been used to improve the respiratory function of tetraplegic patients in the chronic stage of injury. In this study the investigators aim to evaluate whether electrical stimulation of the abdominal muscles can assist the process of weaning from mechanical ventilation in acute ventilator dependent spinal cord injured patients.

DETAILED DESCRIPTION:
Purpose:

The principal aim of this study is to evaluate the feasibility of using Abdominal Functional Electrical Stimulation (AFES) to assist weaning from mechanical ventilator in acute ventilator dependent tetraplegic subjects.

Participants:

10 ventilator dependent tetraplegic participants in the acute stage of injury will be recruited while inpatients at the Queen Elizabeth National Spinal Injuries Unit (QENSIU), Southern General Hospital, Glasgow. The participants will be matched for injury level, age (+/5 years) and sex with a control obtained from historic records of previous patients in the QENSIU.

Experimental Procedures:

Each participant will take part in daily AFES-assisted Weaning sessions (5 times per week) during alternative weeks. Progress will be monitored during weekly Assessment sessions. The total duration of participation is 8 weeks.

AFES-assisted Weaning sessions:

The aim of the weaning sessions is to strengthen the abdominal muscles and to provide support for ventilator free breathing.

The participant will receive AFES training once per day for a predetermined time (see below), 5 days per week. Before the study begins and at the end of each week an assessment session will be conducted.

AFES training sessions will continue throughout even if the patient is successfully weaned before the end of the 8 week period. All procedures will be carried out at the participant's bedside and during all procedures a clinician and the participant's nurse will be present.

The duration of AFES training will initially be 20 minutes/day. This will be increased to 30 minutes in week 3 and to 40 minutes during weeks 5 and 7. While the participant is still not able to breathe independently of the ventilator, AFES will be applied while the participant is connected to the ventilator. As weaning progresses, Spontaneous Breathing Trials (SBTs) will begin and AFES will be applied with the participant disconnected from the ventilator. While the participant is off the ventilator their oxygen saturation level (SaPO2) will be monitored and recorded every minute. Participant will be immediately reconnected to the ventilator if their SaPO2 falls below a clinically critical value of 92%.

Assessment sessions:

An initial assessment session will be conducted on day 1 of the study to provide a baseline measure of the participant's respiratory function. Assessment sessions will then be conducted once per week to assess weaning progress. The assessment sessions will be augmented with a period of AFES training to ensure that the prescribed period of AFES is achieved (see above).

During the assessment sessions the participant's respiratory function (Secondary Outcome Measures) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Acute spinal cord injured tetraplegic patients (patients with a new spinal cord injury) who are inpatients at the Queen Elizabeth National Spinal Injuries Unit (QENSIU), Southern General Hospital, Glasgow;
* Reduced respiratory function requiring mechanical ventilation;
* Good visual response to surface abdominal stimulation, suggesting that lower motor neurons are intact.

Exclusion Criteria:

* Female subjects who are pregnant;
* Significant history of autonomic dysreflexia;
* No visual response to surface abdominal stimulation, suggesting that lower motor neurons are not intact.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to wean from mechanical ventilation | Assessed once per patient
  Time from initial ventilation to achieve 7 days of ventilator free breathing.

SECONDARY OUTCOMES:
Unassisted breathing vital capacity | Up to 8 weeks
  The participant will be asked to breathe without ventilator support. Vital capacity (total lung capacity, VC) will be measured.
AFES assisted breathing tidal volume | Up to 8 weeks
  The participant will be asked to breathe on their own without the support of the ventilator, but with the assistance of abdominal FES. During this time tidal volume will be recorded.
AFES assisted breathing vital capacity | Up to 8 weeks
  The participant will be asked to breathe on their own without the support of the ventilator, but with the assistance of abdominal FES. During this time vital capacity will be recorded.
Unassisted breathing tidal volume | Up to 8 weeks
  The participant will be asked to breathe without ventilator support. Tidal volume (amount of air inhaled and exhaled during a breath, VT) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gollee, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

REFERENCES:
- [Background] McLachlan AJ, McLean AN, Allan DB, Gollee H. Changes in pulmonary function measures following a passive abdominal functional electrical stimulation training program. J Spinal Cord Med. 2013 Mar;36(2):97-103. doi: 10.1179/2045772312Y.0000000031. PMID 23809523
- [Background] Gollee H, Hunt KJ, Allan DB, Fraser MH, McLean AN. Automatic electrical stimulation of abdominal wall muscles increases tidal volume and cough peak flow in tetraplegia. Technol Health Care. 2008;16(4):273-81. PMID 18776604
- [Background] Gollee H, Hunt KJ, Allan DB, Fraser MH, McLean AN. A control system for automatic electrical stimulation of abdominal muscles to assist respiratory function in tetraplegia. Med Eng Phys. 2007 Sep;29(7):799-807. doi: 10.1016/j.medengphy.2006.08.007. Epub 2006 Oct 10. PMID 17035064
- [Background] Lee BB, Boswell-Ruys C, Butler JE, Gandevia SC. Surface functional electrical stimulation of the abdominal muscles to enhance cough and assist tracheostomy decannulation after high-level spinal cord injury. J Spinal Cord Med. 2008;31(1):78-82. doi: 10.1080/10790268.2008.11753985. PMID 18533416
- [Derived] McCaughey EJ, Berry HR, McLean AN, Allan DB, Gollee H. Abdominal Functional Electrical Stimulation to Assist Ventilator Weaning in Acute Tetraplegia: A Cohort Study. PLoS One. 2015 Jun 5;10(6):e0128589. doi: 10.1371/journal.pone.0128589. eCollection 2015. PMID 26047468